CLINICAL TRIAL: NCT01037634
Title: Oseltamivir Treatment in Children Under One Year of Age With Moderate or Severe Influenza Lower Respiratory Tract Infection - a Clinical and Pharmacokinetic Study
Brief Title: Safety and Efficacy of Oseltamivir in Children Younger Than One Year of Age
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: John Tierney, RN, MPM, RCHSPB
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SEA 022
Record Dates: First submitted 2009-12-18; First posted 2009-12-23 (Estimated); Last update posted 2014-08-06 (Estimated); Status verified 2014-08

CONDITIONS: Influenza
Keywords: Avian Influenza; H1N1 Influenza; Seasonal Influenza
MeSH Terms: conditions — Influenza, Human; Influenza in Birds; Orthomyxoviridae Infections | interventions — Oseltamivir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oseltamivir (Experimental): Participants will receive Oseltamivir to treat influenza.
  Interventions: Drug: Oseltamivir

INTERVENTIONS:
Drug: Oseltamivir — 3 mg/kg given orally for 5 days for seasonal influenza, 7 days for 2009 H1N1 influenza (in Vietnam only), or 10 days for avian influenza, for children whose renal function is greater than or equal to 30 mL/min/1.73m2
  Other Names: Tamiflu

SUMMARY:
Currently, there is no standard treatment for influenza with related lower respiratory tract infection (LRTI) in children younger than one year of age, even though influenza related LRTI is a potentially fatal illness in these children. This study will test a medicine for influenza in children younger than one year of age to see if it is safe and effective.

DETAILED DESCRIPTION:
Influenza-related lower respiratory tract infection (LRTI) can cause serious illness or death in children younger than a year old. Only four medications are registered to treat influenza, and these do not have detailed recommendations for treating children younger than one year of age. One of these medications, oseltamivir, has no official recommendation for usage in children younger than one year of age, but it may be the best treatment for certain strains of influenza. A small number of children younger than one year of age have received oseltamivir in several countries with good clinical outcomes and apparently good tolerability. This study will test oseltamivir in children younger than one year of age to see if it is safe and effective.

Children younger than one year of age with influenza will be recruited for this study. Participants will receive the usual care for influenza with the addition of oseltamivir. Oseltamivir will be given orally for 5 days to children with human influenza, 7 days to children with H1N1 influenza in Vietnam, and 10 days to children with avian influenza. Participants will need to remain in the hospital between 5 and 12 days, depending on their illnesses.

Study assessments will be performed daily for 14 days with follow-up examinations occurring 1 to 2 weeks, 6 months, and 12 months after study entry. These assessments will include normal tests for children with influenza, such as blood tests and chest x-rays, but additional blood and nose, throat, and mouth samples will be collected for the study. Participants on a breathing machine will give lung samples.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signed by a parent or legal guardian
* Younger than 12 months of age when first seen with a lower respiratory tract infection (LRTI)
* LRTI must be moderate or severe and influenza must be virologically proven by a respiratory specimen
* History of fever within 14 days prior to presentation (although fever at presentation is not required) plus any two of the following: cough, difficulty breathing or shortness of breath, increased respiratory rate for current age, intercostal recession, use of accessory muscles, nasal flare or grunting, crepitations with or without wheezing, a consistent abnormal chest x-ray (e.g., new infiltrate, hyperinflation)
* Virological evidence of influenza on any one of the tests specified in the protocol

Exclusion Criteria for Children with Non-Avian Influenza:

* Known allergy to oseltamivir

Additional Exclusion Criteria for Children with Non-Avian Influenza:

* Illness duration greater than 14 days on the day of hospital admission
* Creatinine clearance less than 10 mL/min/1.73m2, including a requirement for dialysis or hemofiltration

Ages: 1 Month to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2010-03; Primary Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
Viral clearance of human influenza on a nose and throat swab, assessed by reverse transcriptase polymerase chain reaction (RT PCR) | Measured on Day 5
Viral clearance of H1N1 swine influenza, version found in Vietnam only, on a nose and throat swab, assessed by RT PCR | Measured on Day 7
Viral clearance of avian influenza on a nose and throat swab, assessed by RT PCR | Measured on Day 10

SECONDARY OUTCOMES:
Time to viral clearance on a throat and nose swab, assessed by RT PCR | Measured over 14 days
The time to no detectable influenza virus by culture for the throat and nose swabs | Measured over 14 days
Change in viral load (by log10 copies/mL) over time for all virological samples, with a lower limit of detection of 1,000 copies/mL | Measured over 14 days
Viral susceptibility of cultured influenza virus to antiviral drugs, assessed by genotypical and phenotypical analyses | Measured at baseline and post-treatment
Time to fever clearance | Measured over 14 days
In-hospital mortality and mortality by follow-up | Measured over one year
Time to death | Measured at study completion
Time to trans-cutaneous O2 saturation of greater than or equal to 95% on room air | Measured at study completion
Clinical course: pneumothorax, encephalitis/encephalopathy | Measured at study completion
Number of days in hospital | Measured at study completion
Number of days ventilated | Measured at study completion
Documented serious adverse events (SAEs) and relationships to oseltamivir | Measured at study completion
Adverse events (AEs) leading to drug withdrawal | Measured at study completion
Grade 3 and 4 clinical and laboratory AEs that are probably or definitely related to oseltamivir | Measured at study completion
Skin rashes of any grade | Measured at study completion
Changes in hematological and biochemical parameters over time | Measured at study completion
Pharmacokinetic endpoints, including maximum concentration (Cmax), time of Cmax (Tmax), steady state minimum concentration (Cmin), area under the curve (AUC), and volume of distribution | Measured at baseline, Days 1 to 4, Day 7, and Day 9

CONTACTS AND LOCATIONS:
Overall Officials: Bob Taylor, MD, Principal Investigator — Mahidol Oxford University Research

REFERENCES:
- [Background] Broor S, Parveen S, Bharaj P, Prasad VS, Srinivasulu KN, Sumanth KM, Kapoor SK, Fowler K, Sullender WM. A prospective three-year cohort study of the epidemiology and virology of acute respiratory infections of children in rural India. PLoS One. 2007 Jun 6;2(6):e491. doi: 10.1371/journal.pone.0000491. PMID 17551572
- [Background] American Academy of Pediatrics Committee on Infectious Diseases. Antiviral therapy and prophylaxis for influenza in children. Pediatrics. 2007 Apr;119(4):852-60. doi: 10.1542/peds.2007-0224. PMID 17403862
- [Background] Ferraris O, Lina B. Mutations of neuraminidase implicated in neuraminidase inhibitors resistance. J Clin Virol. 2008 Jan;41(1):13-9. doi: 10.1016/j.jcv.2007.10.020. Epub 2007 Dec 11. PMID 18055254